CLINICAL TRIAL: NCT06182449
Title: Feasibility, Acceptability and Effects of Virtual Reality Distraction for Management of Stress in Mothers Expressing Their Maternal Milk (VR-MOM)
Brief Title: Virtual Reality Distraction for Maternal Milk Expression (PILOT)
Acronym: VR-MOM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Sylvie Le May, Principal Investigator, St. Justine's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VR-MOM-PILOT
Record Dates: First submitted 2023-08-17; First posted 2023-12-27 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Anxiety; Milk Expression, Breast; Breast Milk Collection
MeSH Terms: conditions — Anxiety Disorders; Breast Milk Expression | interventions — AIEOP acute lymphoblastic leukemia protocol

STUDY DESIGN:
Intervention Model Description: The objective is to recruit 20 mothers of premature newborns. This will correspond to a total sample of 40 participants as they will be their own control. We will recruit 50% more mothers (10) to compensate for the usually high attrition or rejection rate for this population, thus a total sample of 30 mothers.
  In addition, allocation to either control or intervention will be randomized at first then switched at the crossover period. However, there will be no washout period between sequences.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Distraction (Experimental): Use of virtual reality (VR) during maternal milk expression.
  Interventions: Device: Virtual Reality Distraction
- Standard Treatment (Active Comparator): Mothers will express their maternal milk in a private room in the NICU with their baby or a photo of the baby.
  Interventions: Other: Standard Protocol

INTERVENTIONS:
Device: Virtual Reality Distraction — In a private NICU room, mothers will wear a head-mounted VR device when they will initiate the expression of their maternal milk. The video within the VR system will provide a calm forest environment with waterfalls, animals, and birdsong (INSPIRE® Program). The baby may or may not be present in the room during the intervention. This will be documented.
  Arms: Virtual Reality Distraction
Other: Standard Protocol — Mothers will express their maternal milk in a private room in the NICU with their baby or a photo of the baby. Use of any co-interventions for anxiety management (e.g. music) durign this sequence will be documented.
  Arms: Standard Treatment

SUMMARY:
Background In neonatal intensive care units (NICUs), mothers are encouraged to express their milk using an electric breast pump. This practice is promoted by nurses and neonatologists due to its beneficial outcomes for newborns. Compared to newborns exclusively fed commercial infant formula, preterm newborns fed breast milk (BM) are less likely to suffer from necrotizing enterocolitis and late-onset sepsis. However, the discomfort associated with using an electrical pump may discourage its use, and almost all mothers start expressing their BM after a premature birth but many stop after a few weeks due to fatigue and stress. Therefore, virtual reality (VR), an immersive experience, seems to be an interesting option as it would provide a relaxing environment and distract mothers of newborns in NICU from the stress and discomfort experienced in order to promote breast milk expression.

Aim

The aim of this within-subject, pilot clinical trial is to assess the feasibility, acceptability, and preliminary effects of VR on stress, discomfort, and volume of expressed milk in mothers of preterm newborns.

Methods

Design:

Within-subject, randomized pilot clinical trial in which participants are their own control.

Setting and sample:

Level 3 neonatal intensive care unit (NICU) at a Montreal pediatric teaching university center. Newborns under 29 weeks of age were chose to ensure that newborns would be admitted and remain in the NICU. The objective is to recruit 20 mothers of premature newborns. This will correspond to a total sample of 40 participants as they will be their own control. There will be 50% more mothers recruited (10) to compensate for the usually high attrition or rejection rate for this population, thus a total sample of 30 mothers. Healthcare professionals (nurses and doctors) providing care to participating mothers will be asked to fill a questionnaire on the feasibility of the VR intervention.

Randomization and exposure to the interventions:

The sequence of exposure to VR will be randomized, not the participants: sequence of 2 days with VR and 2 days without VR. The study will take place over the course of one week. Participating mothers will either be exposed to VR for a minimum of 2 sessions of 30 minutes/day for two days and the following two days to the control intervention or the opposite.

DETAILED DESCRIPTION:
In neonatal intensive care units (NICUs), mothers are encouraged to express their milk using an electric breast pump. The milk is then fed to the premature newborns by a feeding tube until they are stable and mature enough to feed at the breast or by bottle. This practice is promoted by nurses and neonatologists due to its beneficial outcomes for newborns. Compared to newborns exclusively fed commercial infant formula, preterm newborns fed breast milk (BM) are less likely to suffer from necrotizing enterocolitis and late-onset sepsis. In addition, preterm births are often associated with multiple stressors (C-section, separation from the newborn). However, the discomfort associated with using an electrical pump may discourage its use (noise, uncomfortable sensations in the breasts). Overall, almost all mothers start expressing their BM after a premature birth but many stop after a few weeks due to fatigue and stress.

Current recommendations for mothers expressing BM in the NICU include regular skin-to-skin contact as well as being at the bedside or looking at the newborn's photo. Although these methods are effective in increasing BM production, they are not used by all mothers in the NICU. It appears that these strategies remind mothers of being separated from their newborn. Using distraction strategies when expressing BM could be a coping mechanism for such feelings.Few distraction interventions aimed at reducing maternal stress during breast milk expression have been identified in the literature. Some studies have examined the effect of music during milk expression in mothers of newborns hospitalized in the NICU. Researchers observed BM volume increase, nutritional value improvement and maternal cortisol level decrease. Furthermore, interventions focused on relaxation techniques for breastfeeding mothers have shown an increase in milk volume and a weight gain in newborns. Therefore, virtual reality (VR), an immersive experience (auditory and visually) seems to be an interesting option as it would provide a relaxing environment and distract mothers of newborns in NICU from the stress and discomfort experienced in order to promote breast milk expression.

Aim

The aim of this within-subject, pilot clinical trial is to assess the feasibility, acceptability, and preliminary effects of VR on stress, discomfort, and volume of expressed milk in mothers of preterm newborns.

Objectives

1. The primary research objectives are to determine:
2. The feasibility (ease of use, maintenance) of VR with nursing and medical staff
3. The mothers' acceptability and satisfaction of VR
4. The preliminary effects of VR on the volume of breast milk expressed by participating mothers.

The secondary objectives of this study are as follows:

1. To evaluate the preliminary effects of VR on stress levels and discomfort among participating mothers
2. The feasibility of the within-subject clinical trial design (participation, recruitment rate, and questionnaires' response rates, ease of the data collection process, etc.)

Methods

Design:

Within-subject, randomized pilot clinical trial in which participants are their own control.

Setting and sample:

Level 3 neonatal intensive care unit (NICU) at a Montreal pediatric teaching university center. Newborns under 29 weeks of age were chosen to ensure that they would be admitted and remain in the NICU.The objective is to recruit 20 mothers of premature newborns. This will correspond to a total sample of 40 participants as they will be their own control. There will be 50% more mothers (10) recruited to compensate for the usually high attrition or rejection rate for this population, thus a total sample of 30 mothers. Healthcare professionals (nurses and doctors) providing care to participating mothers will be asked to fill a questionnaire on the feasibility of the VR intervention.

Randomization and exposure to the interventions : The sequence of exposure to VR will be randomized, not the participants: sequence of 2 days with VR and 2 days without VR in the same week. The study will take place over the course of one week. Participating mothers will either be exposed to VR for a minimum of 2 sessions of 30 minutes/day for two days and the following two days to the control intervention or the opposite. The frequency of VR use will be documented.

Measures of the primary outcomes

Measures of the feasibility of the VR intervention and the design (healthcare professionals related to participants) : Questionnaires consisting of 10 Likert-type questions ranging from 0 (= strongly disagree) to 4 (= strongly agree), to be completed at the end of the study participation period.

Measures of acceptability and satisfaction with the VR intervention (mothers): Mothers' acceptability will be measured using the Treatment Acceptability & Preference (TAP) questionnaire, 10 questions (6 Likert from 0 (= not at all) to 4 (= strongly) and 4 open-ended questions) as well as with the VAS from 0 (= completely unsatisfied) to 10 (= extremely satisfied) for satisfaction.

Volume of milk expressed: Volume (in mL) of maternal milk expressed by the mother via a breast pump after each milk expression session. Volume will be collected by mothers in a diary provided by the NICU.

Virtual reality specifications

Virtual reality (VR) immerses patients both visually and auditorily in an artificial environment. Inside the virtual reality headset, a depiction of a scene or an imaginary place can be visualized. The INSPIRE Therapeutic Virtual Reality program combines elements of relaxation and sensor-guided deep breathing exercises. The user is immersed in a peaceful forest. In order to lift a feather, the participant has to control her breathing and follow the rhythm suggested. The headset and the relaxation program were designed by Paperplane Therapeutics.

Analyses

Means, standard deviations, and confidence intervals for quantitative data. Paired t-tests to compare the results of the two groups (expressed volume and discomfort). Comparisons of stress at the 4 measurement times using Repeated Measures-ANOVAs (intra- and intersubject comparisons, controlling for carry-over effect). Subgroup analyses (gender, breastfeeding experience, gestational age, number of VR sessions) are planned. A significance level of 0.05 will be used, but the purpose of the study is not to determine the efficacy of VR

ELIGIBILITY:
Inclusion Criteria:

1. speak and read French or English
2. have given birth to a premature newborn at 29 weeks or less
3. minimum 18 years old
4. have chosen breastfeeding
5. who are at least in their second week postpartum

Exclusion Criteria:

1. Having a mental health problem or a significant cognitive disorder that prevents them from understanding the purpose of the study
2. Having a diagnosis of epilepsy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
The feasibility of VR with healthcare professionals | To be reported at the end of the study participation period (1 week).
  Assessing the feasibility (ease of use, maintenance) of VR with nursing and medical staff. Questionnaires consisting of 10 Likert-type questions ranging from 0 to 4.
Mothers' acceptability and satisfaction of VR | Mothers' acceptability will be measured at the end of the study participation (1 week).
  Mothers' acceptability will be measured using the Treatment Acceptability & Preference (TAP) questionnaire, 10 questions (6 Likert from 0 to 4 and 4 open-ended questions) as well as with the Visual Analogue Scale (VAS) from 0 (very dissatisfied) to 10 (very satisfied) for satisfaction
Volume of milk expressed in a day | It will be assessed every time mothers express their milk and the diary will be collected at the end of study participation (1 week).
  Volume (in mL) of maternal milk expressed by the mother via a breast pump in a day. Volume will be collected by mothers in a diary provided by the NICU.

SECONDARY OUTCOMES:
Stress | To be completed before the first sequence (On day 1) , immediately after the first sequence (On day 2), before the second sequence (On day 3) and immediately after the second sequence (On day 4) over the maximum study participation of 1 week.
  Level of stress of mothers will be measured at the beginning and end of each two-days-long sequence with a Visual Analogue Scale (VAS) from 0 to 10, and one of the subscales (Relationships with baby and parental role) of the Parental Stressor Scale-Neonatal Intensive Care Unit (PSS-NICU), 11 Likert-type questions, from 1 to 5.
Discomfort during expression | To be measured immediately at the end of each sequence (On day 2 and day 4) over the maximum study participation of 1 week.
  Level of mothers' discomfort measured at the end of each two-days-long sequence, with a Visual Analogue Scale (VAS) from 0 to 10
Rate of participation | It will be reported in percentage at the end of the study time period (approximately 1 year)
  Rate of participants completing all the measures at the end of the study.
Recruitment rate | It will be reported in percentage at the end of the study period (approx 1 year).
  Rate in percentage of participants recruited for the study
Response rate to the questionnaires | It will be reported in percentage at the end of the study period (approx 1 year).
  Rate in percentage of completed questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Le May, PhD, Principal Investigator — St. Justine's Hospital
Locations (1):
- St.Justine's Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Background] Mizuno K, Ueda A. The maturation and coordination of sucking, swallowing, and respiration in preterm infants. J Pediatr. 2003 Jan;142(1):36-40. doi: 10.1067/mpd.2003.mpd0312. PMID 12520252
- [Background] Schanler RJ, Shulman RJ, Lau C. Feeding strategies for premature infants: beneficial outcomes of feeding fortified human milk versus preterm formula. Pediatrics. 1999 Jun;103(6 Pt 1):1150-7. doi: 10.1542/peds.103.6.1150. PMID 10353922
- [Background] Dieterich CM, Felice JP, O'Sullivan E, Rasmussen KM. Breastfeeding and health outcomes for the mother-infant dyad. Pediatr Clin North Am. 2013 Feb;60(1):31-48. doi: 10.1016/j.pcl.2012.09.010. Epub 2012 Nov 3. PMID 23178059
- [Background] Vohr BR, Poindexter BB, Dusick AM, McKinley LT, Wright LL, Langer JC, Poole WK; NICHD Neonatal Research Network. Beneficial effects of breast milk in the neonatal intensive care unit on the developmental outcome of extremely low birth weight infants at 18 months of age. Pediatrics. 2006 Jul;118(1):e115-23. doi: 10.1542/peds.2005-2382. PMID 16818526
- [Background] Vohr BR, Poindexter BB, Dusick AM, McKinley LT, Higgins RD, Langer JC, Poole WK; National Institute of Child Health and Human Development National Research Network. Persistent beneficial effects of breast milk ingested in the neonatal intensive care unit on outcomes of extremely low birth weight infants at 30 months of age. Pediatrics. 2007 Oct;120(4):e953-9. doi: 10.1542/peds.2006-3227. PMID 17908750
- [Background] Isaacs EB, Fischl BR, Quinn BT, Chong WK, Gadian DG, Lucas A. Impact of breast milk on intelligence quotient, brain size, and white matter development. Pediatr Res. 2010 Apr;67(4):357-62. doi: 10.1203/PDR.0b013e3181d026da. PMID 20035247
- [Background] Infant and Young Child Feeding: Model Chapter for Textbooks for Medical Students and Allied Health Professionals. Geneva: World Health Organization; 2009. Available from http://www.ncbi.nlm.nih.gov/books/NBK148965/ PMID 23905206
- [Background] Keith DR, Weaver BS, Vogel RL. The effect of music-based listening interventions on the volume, fat content, and caloric content of breast milk-produced by mothers of premature and critically ill infants. Adv Neonatal Care. 2012 Apr;12(2):112-9. doi: 10.1097/ANC.0b013e31824d9842. PMID 22469966
- [Background] Juncker HG, Naninck EFG, Schipper L, Lucassen PJ, van Goudoever JB, de Rooij SR, Korosi A. Maternal stress in the postpartum period is associated with altered human milk fatty acid composition. Clin Nutr. 2022 Nov;41(11):2517-2528. doi: 10.1016/j.clnu.2022.09.013. Epub 2022 Sep 28. PMID 36223713
- [Background] Tekgunduz SE, Lazoglu M, Nailoglu M, Apay SE, Tekgunduz KS. The Relationship of Preterm, Term, and Post-Term Births to Maternal Stress and Human Milk Cortisol Levels. Breastfeed Med. 2023 Jun;18(6):462-468. doi: 10.1089/bfm.2023.0006. PMID 37335326
- [Background] Hill PD, Aldag JC, Chatterton RT, Zinaman M. Comparison of milk output between mothers of preterm and term infants: the first 6 weeks after birth. J Hum Lact. 2005 Feb;21(1):22-30. doi: 10.1177/0890334404272407. PMID 15681632
- [Background] Morey JA, Gregory K. Nurse-led education mitigates maternal stress and enhances knowledge in the NICU. MCN Am J Matern Child Nurs. 2012 May-Jun;37(3):182-91. doi: 10.1097/NMC.0b013e31824b4549. PMID 22549422
- [Background] Shaw RJ, Bernard RS, Deblois T, Ikuta LM, Ginzburg K, Koopman C. The relationship between acute stress disorder and posttraumatic stress disorder in the neonatal intensive care unit. Psychosomatics. 2009 Mar-Apr;50(2):131-7. doi: 10.1176/appi.psy.50.2.131. PMID 19377021
- [Background] Foligno S, Finocchi A, Brindisi G, Pace A, Amadio P, Dall'Oglio I, Portanova A, Rossi P, Dotta A, Salvatori G. Evaluation of Mother's Stress during Hospitalization Can Influence the Breastfeeding Rate. Experience in Intensive and Non Intensive Departments. Int J Environ Res Public Health. 2020 Feb 18;17(4):1298. doi: 10.3390/ijerph17041298. PMID 32085465
- [Background] Lebel V, Feeley N, Robins S, Stremler R. Factors Influencing Mothers' Quality of Sleep during Their Infants' NICU Hospitalization. Behav Sleep Med. 2022 Sep-Oct;20(5):610-621. doi: 10.1080/15402002.2021.1971985. Epub 2021 Sep 2. PMID 34472406
- [Background] Acuna-Muga J, Ureta-Velasco N, de la Cruz-Bertolo J, Ballesteros-Lopez R, Sanchez-Martinez R, Miranda-Casabona E, Miguel-Trigoso A, Garcia-San Jose L, Pallas-Alonso C. Volume of milk obtained in relation to location and circumstances of expression in mothers of very low birth weight infants. J Hum Lact. 2014 Feb;30(1):41-6. doi: 10.1177/0890334413509140. Epub 2013 Nov 8. PMID 24212300
- [Background] Hurst N, Engebretson J, Mahoney JS. Providing mother's own milk in the context of the NICU: a paradoxical experience. J Hum Lact. 2013 Aug;29(3):366-73. doi: 10.1177/0890334413485640. Epub 2013 May 1. PMID 23635469
- [Background] Dagli E, Celik N. The effect of oxytocin massage and music on breast milk production and anxiety level of the mothers of premature infants who are in the neonatal intensive care unit: A self-controlled trial. Health Care Women Int. 2022 May;43(5):465-478. doi: 10.1080/07399332.2021.1947286. Epub 2021 Jul 20. PMID 34283710
- [Background] Ak J, Lakshmanagowda PB, G C M P, Goturu J. Impact of music therapy on breast milk secretion in mothers of premature newborns. J Clin Diagn Res. 2015 Apr;9(4):CC04-6. doi: 10.7860/JCDR/2015/11642.5776. Epub 2015 Apr 1. PMID 26023551
- [Background] Mohd Shukri NH, Wells J, Eaton S, Mukhtar F, Petelin A, Jenko-Praznikar Z, Fewtrell M. Randomized controlled trial investigating the effects of a breastfeeding relaxation intervention on maternal psychological state, breast milk outcomes, and infant behavior and growth. Am J Clin Nutr. 2019 Jul 1;110(1):121-130. doi: 10.1093/ajcn/nqz033. PMID 31161202
- [Background] Feher SD, Berger LR, Johnson JD, Wilde JB. Increasing breast milk production for premature infants with a relaxation/imagery audiotape. Pediatrics. 1989 Jan;83(1):57-60. PMID 2642620
- [Background] Miles MS, Funk SG, Carlson J. Parental Stressor Scale: neonatal intensive care unit. Nurs Res. 1993 May-Jun;42(3):148-52. PMID 8506163
- [Background] Sidani S, Epstein DR, Bootzin RR, Moritz P, Miranda J. Assessment of preferences for treatment: validation of a measure. Res Nurs Health. 2009 Aug;32(4):419-31. doi: 10.1002/nur.20329. PMID 19434647